CLINICAL TRIAL: NCT01912651
Title: The Role of Antibiotics in Full Thickness Skin Graft Survival for Facial Reconstructive Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey Moyer, Professor of Otolaryngology-Head and Neck Surgery, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00046677
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Facial Defect
Keywords: facial skin wound; facial wound; skin wound; facial defect; reconstructive skin graft
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No antibiotic treatment (No Intervention): Withholding post-operative antibiotics following reconstructive surgery necessitating skin grafting for defects of the face or nose.
- Antibiotics (Experimental): All patients will receive peri-operative antibiotics per standard practice. This consists of a single dose of cefazolin or, in penicillin allergic patients, clindamycin administered at the time of anesthesia administration prior to the surgical incision. In the cohort randomized to receive post-operative antibiotics, the first choice intervention will be oral cephalexin (500 mg, three times daily or four times daily, for one week). In patients who are penicillin or cephalosporin allergic, we will prescribe clindamycin (300 mg, three times daily or four times daily, for one week).
  Interventions: Drug: cephalexin

INTERVENTIONS:
Drug: cephalexin — This consists of a single dose of cefazolin or, in penicillin allergic patients, clindamycin administered at the time of anesthesia administration prior to the surgical incision. In the cohort randomized to receive post-operative antibiotics, the first choice intervention will be oral cephalexin (500 mg, three times daily or four times daily, for one week). In patients who are penicillin or cephalosporin allergic, we will prescribe clindamycin (300 mg, three times daily or four times daily, for one week). Patients will be followed up within 2 to 6 weeks of surgery and outcome measures assessed. Patients will, again, be seen at 6 months and 1 year post-operatively for outcome assessment.
  Arms: Antibiotics

SUMMARY:
Antibiotics are sometimes prescribed to patients who have had reconstructive surgery of wounds on their face using skin grafts. But, it is not yet known whether antibiotics improve the healing of skin grafts and reduce the risk of infections after surgery in these patients. It is known that antibiotics, like all medications, have side-effects although these are rare. This research study is designed to show us whether antibiotics improve wound healing or not, so that we may determine if we should continue using antibiotics even if they have side-effects in some patients.

Our hypothesis is that patients treated with post-operative, systemic antibiotics will demonstrate a statistically significant improvement in the survival of their facial full thickness skin grafts compared to patients who are not treated with systemic antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with a nasal or facial skin/soft tissue defect requiring reconstruction limited to or including a full-thickness skin graft

Exclusion Criteria:

* current or recent (within one week of surgery) systemic antibiotic use, intolerance to both clindamycin and cephalexin, discovery of a persistent cutaneous malignancy at the site of the defect following the reconstructive procedure and previous reconstruction at the site of the skin/soft-tissue defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Graft failure rate | 1 year
  The primary outcomes will be graft failure rate where failure is defined as any tissue loss extending beyond the epithelium.

SECONDARY OUTCOMES:
Percentage surface area of graft failure | 1 year
  The secondary outcomes include the percentage surface area of graft failure, the incidence of post-operative adjunctive procedures related to graft cosmesis and the incidence of revision surgery resulting from graft failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Moyer, MD, Principal Investigator — University of Michigan Otolaryngology
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States